CLINICAL TRIAL: NCT04972279
Title: Phase 1 Clinical Trial to Develop a Personalized Adaptive Text Message Intervention Using Control Systems Engineering Tools to Increase Physical Activity in Early Adulthood
Brief Title: Precision Assignment of Intervention Messages to Promote Physical Activity - Precision AIM
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, David E Conroy, Professor, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00016346
Record Dates: First submitted 2021-07-12; First posted 2021-07-22 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Cardiovascular Risk Factor

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aggressive adaptation strategy (Experimental): Participants receive up to 6 messages/day to support achievement of their behavior change goal. Messages are only delivered outside of a participant-specific Do Not Disturb window (e.g., 11pm-8am). Messages with coordinating images are selected from three content domains: Move More, Sit Less, and Inspirational Quotes Unrelated to Movement within the first month. The decision rule for each participant will be refined on a monthly basis throughout the 6-month study based upon the accumulating data on how each participant is responding to different messages under different conditions.
  Interventions: Behavioral: Digital message (text + image)
- Moderate adaptation strategy (Experimental): Participants receive up to 3 messages/day to support achievement of their behavior change goal. Messages are only delivered outside of a participant-specific Do Not Disturb window (e.g., 11pm-8am). Messages with coordinating images are selected randomly from three content domains: Move More, Sit Less, and Inspirational Quotes Unrelated to Movement within the first month. The decision rule for each participant will be refined on a monthly basis throughout the 6-month study based upon the accumulating data on how each participant is responding to different messages under different conditions.
  Interventions: Behavioral: Digital message (text + image)

INTERVENTIONS:
Behavioral: Digital message (text + image) — Messages can be up to 256 characters of text with an image. "Move more" and "sit less" messages were written to target established cognitive and affective constructs associated with physical activity (e.g., prompts to action plan, guidance for maximizing pleasure by regulating intensity).

SUMMARY:
Our goal is to develop personalized decision rules for selecting the frequency, timing, and content of messages to promote physical activity. The objective of this project is to evaluate the acceptability and feasibility of two strategies for calibrating decision rules used to send those messages. Participants will wear an activity monitor for the collection of PA data and be randomly assigned to one of two adaptive intervention strategies. The decision rule for each participant will be refined on a monthly basis throughout the 6-month study based upon the accumulating data on how each participant is responding to different messages under different conditions. Our hypothesis is that more intensive intervention strategies will offer a better user experience because the resulting treatments will be experienced as more personalized.

ELIGIBILITY:
Inclusion Criteria:

* Participants capable of reading, speaking and understanding English and of giving informed consent.
* Participants between the ages of 18-29 years.
* Participants must be free of visual impairment that would interfere with the receipt of text messages on their phone.
* Participants must be willing to wear a Fitbit Versa 3 almost continually (23.5 hours/day) for a 6- month period of time.
* Participants must own an iPhone or Android smartphone that they would be willing to download the custom Precision AIM and Fitbit app onto and sync with a Fitbit Versa 3.
* Participants interested in setting goals to increase their physical activity levels over the 6-month study.

Exclusion Criteria:

* Participants engaging in 150 or more minutes of moderate- or greater intensity PA /week as assessed by a research grade accelerometer.
* Participants engaged in organized programs with mandated physical activity (e.g., varsity sports, ROTC).
* Participants with contraindications to normal physical activity on the Physical Activity Readiness Questionnaire.
* Participants who require an assistive device for mobility or have any other condition that may limit or prevent participation in moderate-intensity physical activity.
* Participants who are pregnant or planning to become pregnant within the next 6 months.
* Participants with a prior diagnosis of cancer, cardiovascular disease, diabetes or metabolic syndrome.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2022-01-02 (Actual); Primary Completion 2022-12-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Acceptability of messaging at 6 months | 6 months
  Self-reported preference for more, no change or fewer messages/day based on participant exit interviews coded by two blinded research assistants

SECONDARY OUTCOMES:
Change in total physical activity volume from run-in period | Baseline and 6 months
  Actigraph-assessed total activity counts during a 1-week monitoring period at baseline versus end of study
Change in moderate-to-vigorous physical activity duration from run-in period (baseline) to 6 months(baseline) to 6 months | Baseline and 6 months
  Actigraph-assessed min/week of moderate (or higher) physical activity duration during a 1 week monitoring period at baseline versus end of study

CONTACTS AND LOCATIONS:
Overall Officials: David E Conroy, PhD, Principal Investigator — The Pennsylvania State University
Locations (1):
- The Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No